CLINICAL TRIAL: NCT07153887
Title: An Exploratory Clinical Trial of Vebreltinib for the Treatment of Patients With Locally Advanced or Metastatic Clear Cell Sarcoma
Brief Title: Vebreltinib for Advanced or Metastatic CCS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0507
Record Dates: First submitted 2025-07-20; First posted 2025-09-04 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-06

CONDITIONS: Clear Cell Sarcoma (CCS)
Keywords: CCS; MET; Vebreltinib
MeSH Terms: conditions — Sarcoma, Clear Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vebreltinib Arm (Experimental): subjects will receive Vebreltinib (200 mg bid po) , until disease progression, intolerable toxicity, or death. Subjects will undergo MET abnormality testing after enrollment, including MET amplification or MET protein overexpression.
  Interventions: Drug: Vebreltinib
- External reference arm (Other): Subjects diagnosed with CCS and met the inclusion criteria but refused to enter Cohort1 will receive the standard treatment decided by investigators.
  Interventions: Other: Standard medical treatment

INTERVENTIONS:
Drug: Vebreltinib — Vebreltinib： Oral capsule formulation, specification: 100 mg/capsule. Subjects will start medication after enrollment, 200 mg bid po, until disease progression, intolerable toxicity, or death.
  If disease progression is observed in the first evaluation (2 months after the first administration), if the investigator deems it possible to continue benefiting from targeted therapy, targeted therapy combined with best supportive care can be continued until the second evaluation (4 months).
  Other Names: BoRuiTiNi
  Arms: Vebreltinib Arm
Other: Standard medical treatment — standard treatment like chemotherapy, PD1, Anlotinib……
  Arms: External reference arm

SUMMARY:
This is a prospective, cohort, multicenter study. Cohort 1 is treatment group. All eligible subjects will receive Vebreltinib (200 mg bid po) after signing the informed consent and meeting the inclusion/exclusion criteria, until disease progression, intolerable toxicity, or death. Subjects will undergo MET abnormality testing after enrollment, including MET amplification or MET protein overexpression.

Cohort 2 is external reference group. Subjects diagnosed with CCS and met the inclusion criteria but refused to enter Cohort1 will receive the standard treatment decided by investigators. These subjects will receive follow-up. The efficacy and safety data will be collected.

Imaging evaluation will be performed using RECIST v1.1, with CT or MR plain scans every two months (±7 days) until disease recurrence or death.

During the study, subjects will receive safety follow-up, and survival follow-up will be conducted every two months after treatment, which can be done by telephone interview for approximately 3 years after treatment ends.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥12 years old, male or female;
* ECOG PS score 0-2;
* Histopathologically confirmed unresectable locally advanced or metastatic clear cell sarcoma;
* Previous surgery, radiotherapy, or chemotherapy is allowed; patients who have used PD1/PDL1 for 4 months without effect are allowed to continue using the same PD1/PDL1 drug;
* At least 1 measurable lesion according to RECIST1.1 criteria;
* Normal function of major organs, meeting the following criteria within 7 days before treatment:① Hematology examination criteria must be met (without blood transfusion or blood products, and without correction by G-CSF or other hematopoietic stimulating factors within 14 days):a) Hemoglobin (HB) ≥90g/L; b) Absolute neutrophil count (ANC) ≥1.5×10⁹/L; c) Platelets (PLT) ≥100×10⁹/L; ② Biochemical examination must meet the following criteria: a) Total bilirubin (TBIL) ≤1.5× upper limit of normal (ULN); b) Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×ULN, and if with liver metastasis，ALT and AST ≤5×ULN; c) Serum creatinine (Cr) ≤1.5×ULN or creatinine clearance (CCr) ≥60ml/min; ③ Urine protein <2+, and 24h urine protein quantitation shows protein ≤1g; ④ Coagulation function: INR <2.0 and APTT ≤1.5×ULN ⑤ Doppler ultrasound assessment: Left ventricular ejection fraction (LVEF) ≥ lower limit of normal (60%) ⑥ Thyroid function: TSH ≤ upper limit of normal (ULN); if abnormal, T3 and T4 levels should be considered, and subjects can be enrolled if T3 and T4 levels are normal;
* Male or female of childbearing potential agree to use reliable contraception during treatment and for at least 12 months after the last study drug administration.
* Consent to sign the informed consent form, good compliance, and cooperation with follow-up.

Exclusion Criteria:

* Previous treatment with class Ib MET inhibitors or cabozantinib;
* Clear cell sarcoma with only bone lesions and no soft tissue mass formation;
* Receiving other antitumor treatments within 4 weeks before enrollment, including systemic therapy, radiotherapy, major surgery, or participating in other clinical trials;
* Patients who have not recovered from adverse events caused by previous treatments to NCI-CTCAE (5.0) ≤1 grade, excluding alopecia;
* Subjects with significant bleeding risk determined by the investigator, including but not limited to: 1) Imaging shows that the tumor has invaded important blood vessels or the investigator judges that the tumor is very likely to invade important blood vessels during the subsequent study period, causing fatal massive hemorrhage, or with large vein (iliac vein, inferior vena cava, pulmonary vein, superior vena cava) tumor thrombus formation, or a history of aneurysm with possible rupture; 2) Receiving major surgery or having obvious traumatic injury within 4 weeks before enrollment, or any bleeding or bleeding event ≥NCI-CTCAE grade 3, or any unhealed wound, ulcer, or fracture; 3) Hereditary or acquired bleeding and thrombotic tendencies, such as hemophilia, coagulation disorders, thrombocytopenia, hypersplenism, etc.; 4) Coagulation function abnormalities (INR >1.5 or prothrombin time (PT) >ULN+4 seconds or APTT >1.5 ULN), with bleeding tendency, or receiving thrombolytic or anticoagulant therapy; 5) Patients receiving anticoagulants or vitamin K antagonists such as warfarin, heparin, or their analogs;Note: Under the premise that the international normalized ratio (INR) ≤1.5, low-dose heparin (adult daily dose 0.6×10⁴-1.2×10⁴ U) or low-dose aspirin (daily dose ≤100 mg) is allowed for prophylactic purposes;
* Presence of the following diseases or complications: 1) History of hypertension that cannot be well controlled with 1-2 antihypertensive drugs (systolic blood pressure ≥150mmHg or diastolic blood pressure ≥100mmHg); 2) Poorly controlled diabetes (fasting blood glucose >10mmol/L); 3) Significant cardiovascular damage including but not limited to: unstable angina, myocardial ischemia or infarction, ≥grade 2 congestive heart failure (New York Heart Association (NYHA) classification); history of arterial/venous thromboembolic events within 6 months, such as cerebrovascular accident (including transient ischemic attack), deep vein thrombosis, and pulmonary embolism; 4) Grade I or above sinus bradycardia; or second-degree or above atrioventricular block, or sinus arrest (except with pacemaker); arrhythmia (including QTc ≥480ms); need to take drugs that can prolong QTc. 5) Liver cirrhosis, decompensated liver disease, active hepatitis, or chronic hepatitis requiring antiviral therapy; 6) Urinalysis showing proteinuri≥++, confirmed by 24-hour urine protein quantification > 1.0 g; 7）Renal failure requiring hemodialysis or peritoneal dialysis; 8）History of immunodeficiency, including HIV positivity or other acquired/congenital immunodeficiency diseases, history of organ transplantation or hematopoietic stem cell transplantation, or receiving systemic corticosteroid therapy or any other form of immunosuppressive therapy within 2 weeks before enrollment;Note: In the absence of active autoimmune diseases, inhaled or topical steroids and adrenal cortical hormones at a dose > 10 mg/day prednisone equivalent are allowed, adrenal cortical hormone replacement therapy with a dose not exceeding 10 mg/day prednisone equivalent is allowed, and glucocorticoids are allowed as prophylactic agents for hypersensitivity reactions (such as prophylaxis before docetaxel administration); 9）Active or uncontrolled severe infection (≥ CTC AE grade 2 infection) within 4 weeks before enrollment; 10）Central nervous system metastases confirmed by imaging; 11) History of other malignant tumors within the past 5 years, excluding cured cervical in-situ carcinoma, cutaneous basal cell carcinoma, cutaneous squamous cell carcinoma, and superficial bladder tumors; 12) History of psychoactive substance abuse without abstinence or mental disorders; 13) Receiving ascites/pleural effusion drainage within 2 months before enrollment, or having uncontrolled pericardial effusion, pleural effusion, or ascites; 14) Complications of pulmonary fibrosis or interstitial pneumonia, or severe chronic obstructive pulmonary disease; 15) Severe gastrointestinal diseases, such as gastric perforation, active peptic ulcer, etc.
* Concomitant Medications: 1) Requirement to use strong CYP3A inhibitors (e.g., itraconazole, telithromycin, clarithromycin, ritonavir, etc.) or moderate CYP3A inhibitors (e.g., ciprofloxacin) during the study; 2）Requirement to use strong CYP3A inducers (e.g., phenobarbital, phenytoin sodium, rifampicin, carbamazepine, etc.) or moderate CYP3A inducers during the study; 3）Requirement to take traditional Chinese medicine, especially those with antitumor activity, during the study.
* Others: 1）Anticipated use of any form of systemic or local antitumor therapy during the study; 2）Concomitant diseases or other conditions determined by the investigator to pose a serious risk to the patient's safety, potentially confound study results, or affect the patient's ability to complete the study, such as a gastrointestinal history that may affect oral drug absorption. 3）Subjects with multiple factors affecting oral drug administration (such as inability to swallow, chronic diarrhea, intestinal obstruction, etc.); 4）Allergy to the drugs in this study; 5）Administration of live vaccines within 30 days before enrollment. Live vaccines include but are not limited to: measles, mumps, rubella, varicella/zoster (chickenpox), yellow fever, rabies, Bacille Calmette-Guérin (BCG), typhoid vaccine, etc.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2026-07-15 (Estimated); Study Completion 2027-07-15 (Estimated)

PRIMARY OUTCOMES:
ORR | up to 24 months
  Objective response rate. ORR is defined as the proportion of patients who achieve partial response (PR), or complete response (CR) among all patients.

SECONDARY OUTCOMES:
DCR | up to 24 months
  DCR is defined as the proportion of patients who achieve stable disease (SD), partial response (PR), or complete response (CR) among all patients.
PFS | up to 24 months
  Progression-free survival, is defined as the length of time (months) from randomization to any of the following events: any progression of disease based on response evaluation criteria in solid tumors (RECIST) 1.1, or death due to any cause. Progression is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
OS | up to 24 months
  overall survival, is defined as the time (months) from enrollment to death of participant due to any cause. In the case of a patient who still survives at the time of analysis, the date of last contact will be taken as the censoring date.
12m-OSR | up to 12 months
  12-month overall survival rate. OS is defined as the time (months) from enrollment to death of participant due to any cause. In the case of a patient who still survives at the time of analysis, the date of last contact will be taken as the censoring date.
DOR | up to 24 months
  Duration of response, is defined as the time (months) from partial response to progression of disease.
Treatment-related adverse event (TRAE) | up to 24 months
  Numbers of participants with treatment-related adverse events as assessed by CTCAEv5.0

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No